CLINICAL TRIAL: NCT07026214
Title: Feasibility, Acceptability, and Preliminary Efficacy of a Remotely-delivered Health Coaching Intervention for Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: Holden Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Lucas Carr, Principal Investigator, University of Iowa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 202210267
Record Dates: First submitted 2025-05-30; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-06

CONDITIONS: Cancer
Keywords: health coaching; cancer survivorship
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vitalis Cancer Intervention (Experimental): The intervention includes health coaching, health education, and wearable activity monitoring.
  Interventions: Behavioral: Vitalis Cancer

INTERVENTIONS:
Behavioral: Vitalis Cancer — Participants receive five free health coaching sessions with a trained student health coach, access to three health education videos, and a free wrist worn activity monitor to keep track of their physical activity and sleep behaviors.

SUMMARY:
This study aimed to evaluate the feasibility, acceptability, and preliminary efficacy of an 8-week, remotely delivered health coaching intervention designed to improve: 1) targeted psychosocial mechanisms of action (behavioral regulation skills, affective attitudes, health habits, and identity); 2) health behaviors (physical activity, diet, sleep); and 3) cancer-related health outcomes (physical function, anxiety, depression, fatigue, and pain) among young and middle-aged adult cancer survivors.

DETAILED DESCRIPTION:
Almost 17 million Americans today live with cancer. While advances in cancer treatment have resulted in improved survivorship rates, many treatments are associated with negative, long-term side effects including weight gain, physical dysfunction, fatigue, sleep difficulties, and overall reduced quality of life. Consequently, improving quality of survivorship has been identified as an important but understudied area of research. Both the American Cancer Society and the National Comprehensive Cancer Center Network recommend all cancer survivors maintain a healthy lifestyle that includes being physically active, avoiding inactivity, getting adequate sleep, following a healthy eating pattern, and maintaining a healthy weight. Strong evidence suggests engaging in these healthy lifestyle behaviors has been shown to improve cancer-related health outcomes and quality of life. Unfortunately, most cancer survivors do not meet these recommendations. The American Cancer Society and National Academy of Medicine have recommended healthcare providers and health care systems establish comprehensive survivorship programs that follow patients after primary active treatment and include resources that support engaging in healthy lifestyle behaviors . Unfortunately, a lack of trained survivorship care workforce, lack of reimbursement for survivorship programs, and lack of cohesive systems are major barriers to implementing effective lifestyle behavior survivorship care. Therefore, the aims of this study are:

Aim 1: To determine the feasibility (recruitment rate, attrition rate) and acceptability (program satisfaction) of recruiting and delivering an 8-week remotely delivered lifestyle behavior change intervention to adult cancer survivors.

Aim 2: To determine the efficacy of an 8-week remotely delivered lifestyle behavior change intervention on psychosocial mechanisms of action (behavioral regulation skills, habits, identity), health behaviors (physical activity, sedentary behavior, sleep, diet), and cancer-related health outcomes (anxiety, depression, fatigue, pain, physical function, global health) over 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult cancer survivors aged 18-64 years
* 3-60 months post-treatment
* Not meeting recommendations for physical activity, diet, or sleep.
* Express interest in improving at least one health behavior.

Exclusion Criteria:

* Currently receiving cancer treatment
* Metastatic disease
* Pregnancy or plans for pregnancy
* No access to Zoom or a smartphone

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-09-14 (Actual)

PRIMARY OUTCOMES:
Feasibility - Enrollment | From the first day of study recruitment until the date of the last participant to complete the intervention, assessed up to 36 months
  Enrollment rates calculated as percentage of enrolled vs interested participants
Acceptability | Post-intervention (8 weeks)
  Participants self-reported their acceptability with each intervention feature using an Acceptability Survey. Responses were collected using a 5 point likert scale with higher numbers representing greater satisfaction (1=Very disatisfied, 5=Very Satisfied)
Feasibility Adherence rates | From the first day the intervention launched until the date of the last participant to complete the intervention, assessed up to 36 months
  Participate adherence rates to health coaching sessions calculated as sessions attended vs sessions offered
Feasibility- Retention rate | From the first day of study recruitment until the date of the last participant to complete the intervention, assessed up to 36 months
  Retention rate calculated as percentage comparing number enrolled versus number that complete the study

SECONDARY OUTCOMES:
Behavioral Regulation Skills | From enrollment to 8 weeks
  Participant's perceived ability to regulate their physical activity, diet, and sleep behaviors using a six item survey that uses a 5 point Likert scale. Scores will range from 6 (low skills) to 30 (high skills).
Habit formation skills | From enrollment to 8 weeks
  Habit formation was measured with a 3 question survey using a 5 point likert scale. Responses will range from 3 (weak habit) to 15 (strong habit).
Physical activity | Enrollment to 8 weeks
  Minutes per day of moderate intensity physical activity measured for 7 days with a ActivPAL
Diet behavior | From enrollment to 8 weeks
  Measured with the Automated Self-Administered Dietary Assessment (ASA24) Tool
Sleep behavior | From enrollment to 8 weeks
  Sleep time and sleep efficiency measured for 7 days with an ActTrust2 actigraph
Global Health | From enrollment to 8 weeks
  Measured with two questions on a 5 point likert scale. Scores will range from 2 (poor) to 10 (excellent)

CONTACTS AND LOCATIONS:
Locations (1):
- Lucas J Carr, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No